CLINICAL TRIAL: NCT03837314
Title: Simpler and Safer Deep Brain Stimulation for Parkinson's Disease
Acronym: SPARKS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: North Bristol NHS Trust (Other)
Collaborators: Bioinduction (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3174
Record Dates: First submitted 2015-04-16; First posted 2019-02-12 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deep Brain Stimulation; Neuromodulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Deep Brain stimulation using a novel device. Bioinduction "Picostim" Deep Brain Stimulation system
  Interventions: Device: Bioinduction "Picostim" Deep Brain Stimulation system

INTERVENTIONS:
Device: Bioinduction "Picostim" Deep Brain Stimulation system — Neurostimulation of the subthalamic nucleus region.

SUMMARY:
The aim is to improve availability and acceptability of deep brain stimulation (DBS) for the treatment of Parkinson by shortening and simplifying the implantation procedure, thereby reducing time in surgery, complexity, post-surgery complications and cost, and increasing patient satisfaction.

To facilitate the shortening and simplifying of the implantation procedure, a miniaturised skull-mounted DBS device (Picostim) has been developed which is optimised to generate waveforms needed for stimulation of the subthalamic nucleus (STN) and STN region, employing a unique method of controlling stimulation current. The planned study is a single centre, open label, non-randomised design with the primary objective of showing similarity in control of motor symptoms for the Picostim device compared with previously published data for existing DBS devices.

DETAILED DESCRIPTION:
High-frequency DBS of the STN and STN region is an established treatment for moderate to advanced Parkinson with motor fluctuations, reducing motor symptoms in late stage levodopa responsive patients, who are not adequately controlled by optimal medical therapy alone. However, DBS is presently employed in less than 2% of Parkinson patients. Although a proportion of Parkinson patients are for various reasons not suitable for DBS, currently there is a significant under-utilisation of this approach and in part this is due to perceived surgical risk. Other limitations to adoption are availability of surgeons and infrastructure, particularly outside the USA, and expense.

The objective of this project is to collect and assess safety data for a new DBS device for treatment of Parkinson and validate a new surgical technique employing a skull mounted device. The device, called Picostim, is highly miniaturised and optimised for Parkinson, with current controlled outputs and a rechargeable battery. In typical use, an inductive recharge is required once per week for one hour and service-life is projected to be 17 years. This project aims to advance the technology of DBS so that it is possible to treat a greater proportion of patients more easily, by shortening and simplifying procedures thereby reducing surgical time, complexity and cost, while increasing patient satisfaction and quality of life. Up to 25 patients will receive the Picostim implantation and will be followed up over a one-year period.

This pilot study will be sufficient to make an application for a CE mark in Europe and should inform future studies that are envisaged to be required to prepare an FDA pre-market application.

ELIGIBILITY:
Inclusion criteria:

* Patients who report motor symptoms of Parkinson for at least 4 years;
* Patients eligible for DBS Surgery;
* Receiving stable medical therapy for 30 days or longer before screening assessments - as reported by the patient;
* Males and females aged 21 years or older;
* Be willing and able to comply with all visits and study related procedures (e.g., using the remote control, charging systems and completing the motor diary);
* Understands the study requirements and the treatment procedures and is able to provide written informed consent;
* Females of child-bearing potential must have a negative pregnancy test at study entry and report using an effective method of contraception;

Exclusion criteria:

* Atypical Parkinsonian (Parkinson-plus) syndromes;
* Any prior movement disorder treatments that involved intracranial surgery or device implantation;
* Presence of or planned implant of any other active implanted device;
* Surgical contraindications (such as issues preventing safe anaesthesia);
* Contraindications for MRI scanning (such as presence of metal in the body which means scanning may be harmful);
* Active alcohol or drug abuse;
* Dementia or any neuropsychological condition or finding that would contraindicate DBS surgery. Mattis DRS-2 AEMSS of 6 or less;
* Previous brain surgery likely to interfere with DBS implant;
* Frequent falls when on adequate medication therapy in an "on" state, in the opinion of the PI/delegated clinician;
* A past or current psychiatric disturbance that in the opinion of the PI contraindicates DBS surgery;
* Use of anticoagulant medications that cannot be discontinued during perioperative period;
* Clinically problematic dopamine dysregulation syndrome in the opinion of the PI;
* Significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with expected survival of less than 5 years;
* Participation in another trial concurrently or within 30 days preceding enrolment, that is deemed to interfere with this trial;
* Females who are pregnant, considering becoming pregnant during the study period, or who are breastfeeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in motor function. | 26 weeks
  Change in the Unified Parkinson's Disease Rating Scale (UPDRS) III score at 26 weeks post implantation with stimulation on without medication compared with baseline assessment (without medication). Standard range is from 0 to 108, lower score is better than higher score
Collection and recording of adverse events | 26 weeks
  Rate and type of adverse events including serious adverse events, procedure-related, device-related, stimulation-related, and other adverse events

SECONDARY OUTCOMES:
Surgical time to complete procedure | 12, 26 and 52 weeks intra-operative post device implantation.
  Surgical time to complete procedure. Range being between 2h and 2 days.
Post-operation complications: % of patients with infections and pain at the implantation site | 12 weeks
  % of patients with infections and pain at the implantation site
Tolerability and satisfaction with the head mounted device on a 1-10 range Patient satisfaction questionnaire | 12, 26 and 52 weeks post device implantation.
  User assessment of the tolerability of the head mounted device and of the device's battery efficiency (length and frequency of charging, ease of use) for up to one year following surgery. Assessed through a 1-10 scale, 1 being the worst outcome, 10 the best outcome
Motor functions assessed through recording of motor fluctuation diary | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in motor fluctuation diary recordings at 12, 26 and 52 weeks post implantation.
Mentation, Behaviour and Mood assessed through standard UPDRS Test (see description) | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in motor functions: Unified Parkinson's Disease Rating Scale (UPDRS) I score at 12, 26 and 52 weeks post implantation. UPDRS I score can vary between 0 and 16, 16 being the worst outcome and 0 the best outcome
Motor and cognitive functions | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in L-dopa equivalent. Medication requirements at 12, 26 and 52 weeks post implantation. Range between 300 mg/day and 2000 mg/day, best outcome is lower consumption (300 mg/day)
Motor and cognitive functions assessed through standard Hoehn and Yahr test (see description) | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in Hoehn and Yahr scores at 12, 26 and 52 weeks post implantation. Scale is between 1 to 5, best outcome being 1, worst outcome being 5
Non-Motor functions assessed through standard Dementia Rating Scale (see description) | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in non-motor symptom scores at 12, 26 and 52 weeks post implantation. Dementia Rating scale 2 (DRS-2) score. Range from 0 to 144, 144 being the best outcome.
Cognitive functions assessed through standard Beck Depression Inventory Test (see description) | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in cognitive function and mood status scores at 12, 26 and 52 weeks post implantation. Beck Depression Inventory score, range from 0 to 63, 0 being the best outcome, 63 being the worst outcome
Quality of life assessed through standard Eq5D questionnaire (see description) | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in quality of life measures at 12, 26 and 52 weeks post implantation. EuroQuality of Life score (Eq5D) score ranging from 5 to 15, 5 being the best outcome, 15 the worst.
Activities in Daily Living assessed through standard UPDRS Test (see description) | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in motor functions: Unified Parkinson's Disease Rating Scale (UPDRS) II on and off stimulation at 12, 26 and 52 weeks post implantation. Scores range from 0 to 52, 0 being the best outcome, 52 the worst outcome
Motor examinations assessed through standard UPDRS Test (see description) | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in motor functions: Unified Parkinson's Disease Rating Scale (UPDRS) III score on medications at 12, 26 and 52 weeks post implantation. Scores range from 0 (best outcome) to 56 (worst outcome)
Complications of Therapy assessed through standard UPDRS Test (see description) | 12, 26 and 52 weeks post device implantation.
  Assessment of change from baseline in motor functions: (Unified Parkinson's Disease Rating Scale) UPDRS IV score at 12, 26 and 52 weeks post implantation. Score range from 0 (best outcome) to 23 (worst outcome)
Safety data assessed through analysis of adverse events occurence | 12, 26 and 52 weeks post device implantation.
  Collection and assessment of adverse events (procedure-related, device-related, stimulation-related, and other adverse events) throughout the trial. % of patients having device-related or procedure related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Whone, PhD, Principal Investigator — North Bristol NHS Trust; Nik Patel, MD, Principal Investigator — North Bristol NHS Trust; Steve Gill, MD, Principal Investigator — North Bristol NHS Trust
Locations (1):
- Bristol Brain Centre, Elgar House, Southmead Hospital, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study site and Sponsor — http://www.nbt.nhs.uk/our-services/a-z-services/functional-neurosurgery
- See also: Study funder — http://www.bioinduction.com/